CLINICAL TRIAL: NCT06236919
Title: E-Emotio Project A Gamified Preventive School-based Paradigm Using Virtual Reality Technologies for Improving Emotional Regulation in Children and Adolescents.
Acronym: e-Emotio
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 31607
Record Dates: First submitted 2024-01-12; First posted 2024-02-01 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Emotional Regulation; Virtual Reality; Anxiety; Depression; Executive Function
MeSH Terms: conditions — Emotional Regulation; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR cognitive training (Experimental): The VR cognitive training group will engage in a subset of six games with adaptive difficulty, designed to target specific cognitive functions.
  Interventions: Behavioral: VR cognitive training
- VR nature-exposure relaxation group (Active Comparator): The control group will be immersed in VR nature-based content and perform relaxation exercises.
  Interventions: Behavioral: VR nature exposure relaxation

INTERVENTIONS:
Behavioral: VR cognitive training — The VR cognitive training group will engage in a subset of six games designed to target specific cognitive functions one game will target cognitive flexibility, requiring participants to switch between different tasks and problem-solving strategies quickly. Another game will focus on planning, asking participants to make a series of decisions to achieve a particular goal. Additionally, the Enhance VR group will also engage in games that target reappraisal strategies, working memory, divided and sustained attention, impulsivity, and processing speed.
  Arms: VR cognitive training
Behavioral: VR nature exposure relaxation — The control group will be immersed in ten different nature-based VR environments (e.g., forests, lakes, beaches, etc.), where they will tailor its content and perform relaxation exercises (deep breathing techniques).
  Arms: VR nature-exposure relaxation group

SUMMARY:
Introduction and Significance: Preventive interventions have been shown to reduce the risk of developing anxiety and depression, making them a critical focus area in mental health promotion for children and adolescents. Enhancing emotion regulation (ER) skills in young people is one approach to preventing anxiety and depression, as ER involves cognitive processes of modifying thoughts and behaviors to manage emotional responses in different contexts. Executive functions (EF), such as cognitive flexibility, working memory, and inhibition, play a crucial role in ER development and regulation in children and adolescents. Recently, immersive virtual reality (IVR) has emerged as a novel tool for improving cognitive training interventions' accessibility and effectiveness. IVR allows users to experience immersive, three-dimensional environments, where they can interact with objects and events in a highly engaging and realistic way. Considering these developments, this study aims to explore the potential benefits of Enhance VR, a gamified IVR program designed to improve ER skills and reduce anxiety and depressive symptoms among children and adolescents.

Methodology: The study will be a longitudinal, parallel, single-blind, randomized controlled pilot trial involving 80 Spanish - or English-speaking participants aged 10 to 16 years old. Participants will be excluded if they have severe psychiatric or neurodevelopmental disorders, physical, motor, or sensory impairments, or a risk of experiencing high cybersickness symptomatology during the VR experience. Participants will be randomly allocated into two groups: an experimental group receiving E-Emotio VR and a control group receiving a placebo-based VR relaxation experience. Both VR interventions will last five weeks, two times a week, for 30 minutes. The experimental group will engage in six games targeting cognitive flexibility, planning, reappraisal strategies, working memory, divided and sustained attention, and processing speed. The control group will be immersed in ten different nature-based VR environments and perform relaxation exercises. Baseline and post-intervention assessments will be conducted using age-adapted validated measures of depressive and anxiety symptoms, ER, executive function (working memory, cognitive flexibility, inhibition, and planning), and attention. Following the intervention, the assessment battery will be re-administered by a blinded assessor, and statistical analyses will be conducted for all the primary and secondary measures assessed before and after the intervention in both groups.

Conclusion: In summary, this study aims to contribute to the development of effective preventive interventions for emotion regulation and mental health symptoms in children and adolescents by promoting ER through gamified VR cognitive training. The study's findings could have significant implications for mental health research, educational and clinical practice. By exploring the potential benefits of VR cognitive training, this research has the potential to inform future studies and clinical interventions aimed at improving young people's mental health and well-being. The gamification of cognitive training interventions could be a powerful tool for increasing engagement and motivation among young people, making them more likely to participate in such interventions.

ELIGIBILITY:
Inclusion Criteria:

* School-aged participants (aged 10 to 16 years old)
* Individuals who provide consent to participate.

Exclusion Criteria:

* A previous diagnosis of severe psychiatric (e.g., maniac, or psychotic symptoms).
* A previous diagnosis of severe psychiatric neurodevelopmental disorders (i.e., severe autism spectrum disorders, intellectual disabilities, etc),
* A previous diagnosis of severe physical, motor, or sensory impairments that could interfere with the examination or the VR program.
* Participants who cannot understand Spanish.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA) | At baseline and after 5 weeks.
  The ERQ-CA comprises 10 items assessing the emotion regulation strategies. Items are rated on a 5-point Likert-type response scale, with a minimum and maximum range of scores from 10-50. Higher scores on each scale indicate greater use of emotion regulation strategies.
Revised Child Anxiety and Depression Scale (RCADS-47) | At baseline
  The Revised Child Anxiety and Depression Scale (RCADS-47) is a 47-item, youth self-report questionnaire that assess Anxiety and Depression symptoms including six subscales: separation anxiety disorder (SAD), social phobia (SP), generalized anxiety disorder (GAD), panic disorder (PD), obsessive compulsive disorder (OCD), and major depressive disorder (MDD). It also yields a Total Anxiety Scale (sum of the 5 anxiety subscales) and a Total Internalizing Scale (sum of all 6 subscales). Items are rated on a 4-point Likert-scale from 0 ("never") to 3 ("always") with a minimum and maximum range of scores from 0-141. Higher scores indicate higher levels of Anxiety and/or Depression.
State-Trait Anxiety Inventory for Children (STAI-C) | At baseline and after 5 weeks.
  The State-Trait Anxiety Inventory for Children (STAI-C) item self-rated scale that assesses the two dimensions of anxiety in children; 1) state anxiety as a temporary emotional condition; 2) and trait anxiety as a relatively stable anxious tendency. This inventory has 40 items, which are answered with an ordinal scale with 4 options (0 to 3, from "almost never" to "always") with a minimum and maximum range of scores from 0-60 in each scale. Higher scores indicate higher levels of Anxiety.
Children's Depression Inventory (CDI) | At baseline and after 5 weeks.
  The Children's Depression Inventory (CDI) is a 27 item self-rated scale that assesses Depression symptoms in children. Each item is answered with a 3-point Likert-scale from 0 "absence of the symptom" to 2 "severe symptom" with a minimum and maximum range of scores from 0-54. Higher scores indicate higher levels or risk of Depression.
Positive and Negative Affect Schedule (PANAS) | At baseline and after 5 weeks.
  The Positive and Negative Affect Schedule is a brief scale of 20 items, with 10 items measuring positive affect (e.g., excited, inspired) and 10 items measuring negative affect (e.g., upset, afraid). Each item is rated on a five-point Likert Scale, ranging from 1 = Very Slightly or Not at all to 5 = Extremely, to measure the extent to which the affect has been experienced in a specified time frame. The scale can be used to measure state affect, dispositional or trait affect, emotional fluctuations throughout a specific period of time, or emotional responses to events.

SECONDARY OUTCOMES:
General Self-Efficacy Scale (GSE) | At baseline and after 5 weeks.
  The General Self-Efficacy Scale (GSE) is a self-report measure of self-efficacy that assesses the stable feeling of personal competence to effectively handle a large variety of stressful situations. This scale comprises 10 items and each item is answered with a 10-point Likert-scale from 1 to 10. This scale has a minimum and maximum range of scores from 10-100. Higher scores indicate more self-efficacy perception.
Ruminative Response Scale (RRS-SF) | At baseline and after 5 weeks.
  The Ruminative Response Scale (RRS-SF) is a self-report measure that describes individual responses to negative emotions describing self and symptom-focused responses to depressed mood. This scale includes 10 items and is rated on a 4-point Likert scale ranging from 1 (never) to 4 (always). The total score ranges from 10 to 40. Higher scores indicate higher degrees of ruminative symptoms.
Child's Report of Parental Behavior Inventory Abbreviated (CRPBI-A) | At baseline and after 5 weeks.
  The 29-item abbreviated form of the questionnaire (CRPBI-A) consists of six scales assessing the following 6 child-rearing styles: communicative, hostile/rejection, controlling, permissive, overprotective, and negligent for both mother and father. This scale is rated on a 3-point Likert scale ranging from 1 (almost never) to 3 (many times).
Behavior Rating Inventory of Executive Function 2 (BRIEF-2) | At baseline and after 5 weeks.
  The BRIEF-2 questionnaire is a test intended for the evaluation of the most everyday, behavioral and observable aspects of the executive functions of children and adolescents between 5 and 18 years old. The questionnaire can be self-reported (BRIEF-" Self-report) answered by family members (BRIEF-2 Family) and by teachers (BRIEF-2 School), who must indicate the frequency with which certain behaviors are problematic.
  It consists of 63 items that are answered with a frequency scale (never, sometimes times, frequently) in a time of approximately 10 minutes, and it evaluates different scales related to executive functions: inhibition, self-monitoring, flexibility, emotional control, initiative, working memory, planning and organization, task supervision and materials organization.
Stroop Color and Word Test (SCWT) | At baseline and after 5 weeks.
  Selective attention, inhibition, and processing speed are measured with the Stroop Color and Word Test (SCWT). Participants are asked to name the color of a series of color patches (Stroop Color Naming), read a series of color words (Stroop Word Reading), and name the color of a series of color words where the word and color do not match (e.g., the word "red" written in blue ink), Stroop Color-Word Interference. Higher scores mean a better outcome.
Trail Making Test A and B (TMT A-B) | At baseline and after 5 weeks.
  The Trail Making Test (TMT) is a freely available, timed, neuropsychological test that involves visual scanning and working memory. The TMT has two parts; the TMT-A (visual scanning and processing speed) and TMT-B (executive functioning and cognitive flexibility). In each test the participant is asked to draw a line between 24 consecutive circles that are randomly arranged on a page. The TMT-A uses all numbers, whereas the TMT-B alternates numbers and letters, requiring the patient to switch between numbers and letters in consecutive order. The TMT is scored by how long it takes to complete the test. The time includes correction of errors prompted by the examiner. If the person cannot complete the test in 5 minutes, the test is discontinued. Higher scores mean a better outcome.
Digit forward and backward span | At baseline and after 5 weeks.
  Digit Span Forward requires the child to repeat numbers in the same order as read aloud by the examiner (auditory attention), and Digit Span Backward requires the child to repeat the numbers in the reverse order of that presented by the examiner (verbal working memory). Every item on Digit Span consists of two trials, each of which is scored 1 or 0 points. Pacing of the item stimuli is critical on Digit Span, as variations in how quickly or slowly they are provided can greatly impact item difficulty. The numbers are read at the rate of one per second, and there are a number of techniques that examiners use to establish an accurate, consistent pace. The Longest Digit Span Forward (LDSF) and Longest Digit Span Backward (LDSB) process scores permit examination of maximum performance on each task relative to the normative sample. Higher scores mean a better outcome.
Wisconsin Card Sorting Test Computer Version 4-Research Edition (WCST:CV4) | At baseline and after 5 weeks.
  The Wisconsin Card Sorting Test (WCST) was created to evaluate the capacity of abstraction, the formation of concepts and the change of cognitive strategies in response to the changes that occur in environmental contingencies. The WCST is used in people from 6,5 years old to 89 and it is made up of 1 set of 64 cards. The cards are composed of a combination of 3 types of attributes or characteristics: shape (triangle, star, cross and circle), color (red, blue, green and yellow) and number (1, 2, 3 or 4 elements). The task is to distribute the cards matching one criterion. When the subject makes 10 consecutive correct answers, it is considered that a category has ended, from then on the classification criterion is changed without prior warning. If you continue classifying the cards with the criteria of the previous category, you will score in perseverative errors.The test ends when the subject completes all 6 series or categories, or when the subject completes 128 trials.
System Usability Scale (SUS) | After 5 weeks.
  The System Usability Scale (SUS) is a self-report measure that evaluates the usability of a wide variety of products and services, including hardware, software, mobile devices, websites and applications. It consists of a 10 item questionnaire that is rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score ranges from 10-50 with higher scores indicating greater levels of usability.
Simulator Sickness Questionnaire (SSQ) | After 5 weeks.
  The Simulator Sickness Questionnaire (SSQ) is a self-report measure that is used to assess cybersickness or adverse symptoms associated with VR. It consists of a 16 item questionnaire that is rated on a 4-point Likert scale ranging from 1 ("no symptoms") to 3 ("severe symptoms"). The total score ranges from 10 to 30 with higher scores indicating higher levels of adverse symptoms.
Visual Analogue Scales (VAS) | After each IVR session (Every session, twice a week, for 5 weeks)
  Visual Analogue Scales (VAS) are psychometric response scales used to measure subjective characteristics or attitudes. The participants have to rate the intensity of their feeling of Immersion and Enjoyment on a scale from 0 (none) - 100 (completely) after the completion of all IVR tasks of each session. Both questions will be asked orally to each participant:
  1. "Rate from 0 to 100 the degree of immersion that you felt inside the virtual environment. With 0 being none and 100 being completely".
  2. "Rate from 0 to 100 how much you liked the virtual environment. With 0 being not at all and 100 being completely".

CONTACTS AND LOCATIONS:
Locations (1):
- UIC Barcelona International University of Catalonia, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No